CLINICAL TRIAL: NCT02586324
Title: Comparison of Two Embryo Culture Media for IVF (in Vitro Fertilization) and ICSI ( Intracytoplasmic Sperm Injection ): Randomized Prospective Study
Brief Title: Comparison of Two Embryo Culture Media for IVF and ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JIMENEZ 2008
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Culture, ICSI, IVF

ARMS (2):
- global medium (Other)
  Interventions: Biological: global medium
- SSM (Experimental)
  Interventions: Biological: SSM

INTERVENTIONS:
Biological: global medium
  Arms: global medium
Biological: SSM
  Arms: SSM

SUMMARY:
In this research, the two media used are Global medium and SSM medium with serum), which are routinely used in the reproduction biology unit. This study simply consists in setting up a methodology to compare these to media. The only constraint placed on patients is to accept randomization for the type of medium used.

ELIGIBILITY:
Inclusion Criteria:

* Any IVF and IVF with ICSI procedure performed in the unit can be included in the study

Exclusion Criteria:

* refusal of patients to be randomized. In this case, the biologist chose the medium to be used and the IVF procedure will not be included in the statistical analysis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Rate of pregnancies and deliveries | Up to 9 months